CLINICAL TRIAL: NCT01356979
Title: Outcome of Patients Who Could Not Have Been Diagnosed by Medical Thoracoscopy
Brief Title: Outcome of Patients Undiagnosed Under Medical Thoracoscopy
Status: Completed | Type: Observational
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Muzaffer Metintas, MD, Prof. in Pulmonary Medicine, Eskisehir Osmangazi University
Other Study IDs: 052011/15
Record Dates: First submitted 2011-05-16; First posted 2011-05-20 (Estimated); Last update posted 2012-09-25 (Estimated); Status verified 2012-09

CONDITIONS: Pleural Diseases
Keywords: Medical thoracoscopy; Pleural effusion; Malignant pleural diseases; Tuberculous pleuritis; Fibrinous pleuritis
MeSH Terms: conditions — Pleural Diseases; Pleural Effusion; Tuberculosis, Pleural

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients underwent medical thoracoscopy: Patients who require medical thoracoscopy for undiagnosed exudative pleural effusion by other clinical or radiological investigations.
  Interventions: Procedure: Medical thoracoscopy

INTERVENTIONS:
Procedure: Medical thoracoscopy — Performing medical thoracoscopy to diagnose pleural diseases after cytological and other investigational tests.
  Other Names: Rigid thoracoscopy for diagnosis of pleural diseases

SUMMARY:
Medical thoracoscopy (MT) under local anaesthetic and mild sedation, an established method in the diagnosis of pleural diseases. MT has an overall diagnostic yield above 90% for malignant pleural diseases and pleural tuberculosis. However, others who are diagnosed as fibrinous pleuritis make confusion in clinicians. Whether these patients are firmly followed or not ? The investigators do not know the answer of this question.

In this study the investigators aimed to investigate the outcome of the patients who are diagnosed as fibrinous pleuritis on MT biopsies.

DETAILED DESCRIPTION:
Medical thoracoscopy (MT) under local anaesthetic and mild sedation, an established method in the diagnosis of pleural diseases with a sensitivity above 90% and specificity of 1000% for malignant pleural diseases and pleural tuberculosis. Except these two groups of patients, in others pleural histopathological diagnosis is defined as "non-specific pleuritis" or "fibrinous pleuritis". Authors say that the natural evolution of these patients is poorly understood. Some of these patients was later established false negative cases for malignant pleural diseases. Clinical guidelines recommend close observation of patients with undiagnosed exudative effusions, although the length and follow-up regime is not defined, yet. In this study the investigators examine the outcome of patients who are diagnosed as fibrinous pleuritis by MT.

ELIGIBILITY:
Inclusion Criteria:

* Undiagnosed exudative pleural effusion
* Under 20 years-old, over 85 years-old
* Followed 2 years at least

Exclusion Criteria:

* Transudative pleural effusion
* Patients who do not accepted medical thoracoscopy.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients with undiagnosed exudative pelural effusion by clinical, radiological or laboratory investigations.
Sampling Method: Probability Sample
Enrollment: 355 (Estimated)
Dates: Start 2002-02; Primary Completion 2009-05 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Accuracy of medical thoracoscopy for patients diagnosed as fibrinous pleuritis. | 2 years
  During 2 years after medical thoracoscopy, the diagnostic sensitivity, specificity, positive predictive value and negative predictive value are determined in the patients diagnosed as fibrinous pleuritis.

SECONDARY OUTCOMES:
To determine the factors which point the false positive diagnosis of fibrinous pleuritis. | 2 years
  The factors predictive of false-negative biopsy results in the patients with a diagnosis of fibrinous pleuritis are determined by using logistic regression analysis .

CONTACTS AND LOCATIONS:
Overall Officials: Muzaffer Metintas, MD, Principal Investigator — ESOGU Medical Faculty Department of Chest Diseases
Locations (1):
- ESOGU Medical Faculty Department of Chest Diseases, Eskişehir, Meselik - Eskisehir, Turkey (Türkiye)